CLINICAL TRIAL: NCT02608489
Title: Clinical Effects and Safety of 3% Diquafosol Ophthalmic Solution for Patients With Dry Eye After Cataract Surgery: A Randomized Controlled Trial
Brief Title: Clinical Effects and Safety of 3% Diquafosol After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jin Kwon Chung, Assistant Professor, Cornea & Refractive Surgery Service, Department of Ophthalmology, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHUH 2013-12-012
Record Dates: First submitted 2015-11-14; First posted 2015-11-18 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — diquafosol; Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diqufosol (Active Comparator): 3% Diquafosol Tetrasodium Ophthalmic Solution
  Interventions: Drug: Diquafosol (Diquas)
- Hyaluronate (Placebo Comparator): 0.1% Sodium Hyaluronate Ophthalmic Solution
  Interventions: Drug: Sodium Hyaluronate (Hyalein)

INTERVENTIONS:
Drug: Diquafosol (Diquas) — Diquafosol group used diquafosol 6 times a day during study period.
  Arms: Diqufosol
Drug: Sodium Hyaluronate (Hyalein) — Hyaluronate group used sodium hyaluronate 6 times a day during study period.
  Arms: Hyaluronate

SUMMARY:
The purpose of this study is determine whether 3% diquafosol and 0.1% sodium hyaluronate are effective and safe in the treatment of patients with dry eye after cataract surgery.

DETAILED DESCRIPTION:
Study group and protocol: This was a prospective open-label randomized study. All patients were given a full explanation of the study, and written informed consent was obtained from all participants. The study protocol adhered to the tenets of the Declaration of Helsinki. The Institutional Review Board and Ethics Committee, Soonchunhyang University Seoul Hospital, approved this study (SCHUH 2013-12-012). Patients were randomly allocated into the diquafosol group (D group) or the hyaluronate group (H group) using a simple unrestricted randomization method by the controller. The D group used 3% diquafosol tetrasodium ophthalmic solution (Diquas®; Santen Pharmaceutical Co., Ltd., Osaka, Japan) six times a day and the H group used 0.1% sodium hyaluronate ophthalmic solution (Hyalein®; Santen Pharmaceutical Co., Ltd., Osaka, Japan) six times a day. Both groups instilled each eye drop from postoperative day 1 to postoperative week 12.

Participants: Consecutive patients aged 20-90 years with bilateral or unilateral cataract undergoing uncomplicated phacoemulsification and intraocular lens (IOL) implantation at Soonchunhyang University Hospital between January 2014 and January 2015 were enrolled. The inclusion criteria were patients with mild to moderate dry eye (level 1 or 2) based on the dry eye severity scale adopted by the Dry Eye Workshop (DEWS) report and who used only artificial tears occasionally1, and patients without or with mild blepharitis.18 The exclusion criteria were presence of any complications after cataract surgery such as cystoid macular edema, patients using any topical eye drops on a regular basis, treatment history of dry eye beyond artificial tears, any ocular surgery within the prior 6 months, contact lens wear, serious ocular surface disease (e.g., Sjögren's syndrome, ocular pemphigoid, conjunctival scarring, chemical injury), lacrimal or eyelid disease (e.g., moderate to severe blepharitis18), use of concomitant medications that could cause dry eye (e.g., antihistamines, antidepressants, decongestants, anticholinergic drugs), and allergy to any of the study medications.

Objective and subjective clinical assessments of dry eye: All patients underwent ophthalmic examinations preoperatively and postoperatively in the order of following : uncorrected distant visual acuity (UDVA) test, an ocular surface disease index (OSDI) questionnaire, Schirmer I test without anesthesia, changes in HOAs after blinking, tear break-up time (TBUT), corneal fluorescein staining, and lissamine green (LG) conjunctival staining. Eyelid and anterior chamber cells were evaluated by slit-lamp biomicroscopy to assess the presence of blepharitis/meibomian gland plugging and intraocular inflammation. Routine postoperative examinations were scheduled for 1 week, 4 weeks, and 12 weeks after surgery.

Efficacy and safety evaluation: To evaluate the efficacy of the two different eye drops, we compared each measurement between the two groups throughout the study period, and at each follow-up, and also compared the patterns of changes in each group to identify which group recovered earlier. we evaluated the safety of the two eye drops, including anterior chamber inflammation and discontinuation of the eye drops due to drug-related discomfort. Patients that had any adverse events or wanted to stop using the eye drops were excluded from the study, but these patients were included in the safety evaluation.

Surgical procedure: A 2.8 mm clear corneal incision was made at the location of the steep corneal astigmatism axis. A standard phacoemulsification technique was used with topical anesthesia with 2% lidocaine. A foldable IOL was implanted into the capsular bag. There was no suture at the corneal incision site. Patients received moxifloxacin (Vigamox; Alcon, Fort Worth, TX), which is a preservative-free formulation, and rimexolone (Vexol; Alcon), which contains 0.01% BAK, four times a day after surgery for 4 weeks.

Statistical analysis: For statistical analysis, UDVA was converted from Snellen into logMAR values. Baseline data were compared between the groups using the Mann-Whitney U-test, Fisher's exact test, and the linear mixed model after adjusting for inter-eye correlations, age, and sex. In addition, another mixed model was used to compare measurement data between the two groups by considering the correlation between both eyes of each patient at each follow-up. To obtain an overall comparison between treatment responses throughout the study period considering the two levels of correlation in subjects and follow-up, a bivariate generalized linear mixed (GLM) model with asymmetric random effects was used. In the last step, a bivariate GLM model was also used to identify the patterns of changes in measured data throughout the study period. The intergroup differences in adverse events were analyzed using Fisher's exact test. SPSS software (version 21, SPSS, Inc., Chicago, IL) was used for all statistical analyses, and P < .05 was taken to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral or unilateral cataract undergoing phacoemulsification and intraocular lens (IOL) implantation at Soonchunhyang University Hospital between January 2014 and January 2015
* Patients with mild to moderate dry eye (level 1 or 2) based on the dry eye severity scale adopted by the Dry Eye Workshop (DEWS) report and who used only artificial tears occasionally

Exclusion Criteria:

* Presence of any complications after cataract surgery such as cystoid macular edema
* Patients using any topical eye drops on a regular basis
* Treatment history of dry eye beyond artificial tears
* Any ocular surgery within the prior 6 months
* Contact lens wear
* Serious ocular surface disease (e.g., Sjögren's syndrome, ocular pemphigoid, conjunctival scarring, chemical injury)
* Eyelid or lacrimal disease
* Use of concomitant medications that could cause dry eye and allergy to any of the study medications

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Kwon Chung, MD, Principal Investigator — Soonchunhyang University Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients aged 20-90 years with bilateral or unilateral cataract undergoing uncomplicated phacoemulsification and intraocular lens (IOL) implantation at Soonchunhyang University Hospital between January 1, 2014 and January 31, 2015 were enrolled.
Period: Overall Study
Arm/Group | Diqufosol | Hyaluronate
Started | 43 | 43
Completed | 30 | 33
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diqufosol | Hyaluronate | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.53 (11.15) | 65.37 (10.02) | 65.45 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 24 | 42
  Male | 12 | 9 | 21
Obstructive Meibomian Gland Dysfunction (MGD) [Number; unit: participants]
  None | 17 | 19 | 36
  Mild | 13 | 14 | 27
Ocular Surface Disease Index ± SD [Mean (Standard Deviation); unit: Scores on a scale] — scale ranges (0-100). Higher values represent a worse outcome.
  Scores on a scale | 22.23 (14.65) | 23.64 (16.62) | 22.96 (15.11)
tear Break-Up Time ± SD [Mean (Standard Deviation); unit: seconds] | 4.88 (2.52) | 4.54 (1.85) | 4.70 (2.06)
Schirmer test ± SD [Mean (Standard Deviation); unit: mm] | 3.52 (4.13) | 3.67 (2.88) | 3.58 (3.31)
Fluorescein staining score ± SD [Mean (Standard Deviation); unit: score] — Instillation of fluorescein in both eyes. After 1 or 2 full blinks, the intensity of staining of both cornea was scored. According to the National Eye Institute (NEI) workshop grading system, the cornea was divided into five sections. The minimum staining score was 0 and the maximum staining score was 15 points (up to 3 points for each section).
  0 : best score (no corneal damage) 15 : worst score (severe corneal damages)
  score | 1.62 (1.77) | 1.77 (1.73) | 1.69 (1.75)
Lissamine green staining score ± SD [Mean (Standard Deviation); unit: score] — Instillation of 1% lissamine green in both eyes. After 1 or 2 full blinks, the intensity of staining of both medial and lateral bulbar conjunctiva was cored. According to the National Eye Institute (NEI) workshop grading system, the conjunctiva was divided into six sections. The minimum staining score was 0 and the maximum staining score was 18 points (up to 3 points for each section).
  0 : best score (no conjunctival damage) 18 : worst score (severe conjunctival damages)
  score | 1.55 (1.19) | 1.94 (1.56) | 1.79 (1.38)
Total High Order Aberration (HOA) changes ± SD [Mean (Standard Deviation); unit: microns] | 0.042 (0.041) | 0.041 (0.048) | 0.041 (0.045)
Uncorrected visual acuity (LogMAR) ± SD [Mean (Standard Deviation); unit: logMAR] | 0.80 (0.52) | 0.77 (0.45) | 0.78 (0.47)
Grade of anterior chamber cells [Mean (Standard Deviation); unit: grade] — Grade ranges (0-4+), Evaluate cells using slit-lamp biomicroscopy. The slit beam should be 1mm x 1mm.
  Grade 0 : < 1 cell in field, Grade 0.5+ : 1-5 cells in field, Grade 1+ : 6-15 cells in field, Grade 2+ : 16-25 cells in fields Grade 3+ : 26-50 cells in field, Grade 4+ : 50+ cells in fields
  grade | 0 (0) | 0 (0) | 0 (0)

OUTCOME MEASURES:

1. Primary Outcome: an Ocular Surface Disease Index (OSDI) Questionnaire That is Related to Dry Eye Severity.
Description: The OSDI questionnaire consists of 12 questions that evaluate subjective symptoms related to dry eye and vision The score ranges were between 0 and 100 scores and the higher scores represent a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Eyes
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 30 | 33
Number analyzed (Eyes) | 45 | 49
scores on a scale
  Baseline | 21.09 (3.86) | 23.00 (2.66)
  Postoperative week 1 | 31.28 (5.49) | 20.31 (4.63)
  Postoperative week 4 | 20.31 (4.63) | 23.00 (3.19)
  Postoperative week 12 | 9.76 (7.95) | 16.92 (13.11)
Statistical Analysis 1: Comparison: Diqufosol vs Hyaluronate; To obtain an overall comparison between treatment responses throughout the study period considering the 2 levels of correlation in subjects and follow-up, a linear mixed model with asymmetric random effects was used; Test type: Superiority or Other; p = 0.221, Mixed Models Analysis
Statistical Analysis 2: Comparison: Diqufosol vs Hyaluronate; Linear mixed model was used to compare measurement data between the 2 groups by considering the correlation between both eyes of each patient at postoperative week 12 follow-up; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis

2. Primary Outcome: Schirmer I Test Without Anesthesia That is Related to Dry Eye Severity.
Description: Schirmer paper strips were placed into the temporal one third of the lower conjunctival sac for 5 min and the wetness on the strips was measured.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 30 | 33
Number analyzed (eyes) | 45 | 49
mm
  Baseline | 3.61 (0.84) | 3.69 (0.58)
  Postoperative week 1 | 2.03 (0.37) | 1.76 (0.25)
  Postoperative week 4 | 3.22 (0.62) | 2.59 (0.43)
  Postoperative week 12 | 4.10 (2.87) | 2.52 (2.08)
Statistical Analysis 1: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.256, Mixed Models Analysis
Statistical Analysis 2: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis

3. Primary Outcome: Changes in HOAs After Blinking That is Related to Dry Eye Severity.
Description: Corneal HOAs and serial measurement of ocular total HOAs were evaluated using a KR-1W wavefront analyzer (Topcon Medical System, Inc., Tokyo, Japan). Serial measurement of total ocular HOAs was measured every second for 10 s after complete blinking in continuous measurement mode. The difference between the fifth and first HOA was used to evaluate the tear film instability.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: eyes
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 30 | 33
Number analyzed (eyes) | 45 | 49
microns
  Baseline | 0.042 (0.010) | 0.041 (0.007)
  Postoperative week 1 | 0.153 (0.057) | 0.260 (0.040)
  Postoperative week 4 | 0.067 (0.029) | 0.074 (0.043)
  Postoperative week 12 | 0.034 (0.040) | 0.039 (0.147)
Statistical Analysis 1: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.080, Mixed Models Analysis
Statistical Analysis 2: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis

4. Primary Outcome: Tear Break-up Time (TBUT) That is Related to Dry Eye Severity.
Description: TBUT was assessed by instillation of a drop of 2% sterile fluorescein into the conjunctival sac and recording the interval between the last complete blink and the first appearance of a dry spot or disruption of the tear film.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 30 | 33
Number analyzed (eyes) | 45 | 49
seconds
  Baseline | 4.98 (0.53) | 4.50 (0.36)
  Postoperative week 1 | 3.50 (1.35) | 3.00 (1.16)
  Postoperative week 4 | 5.64 (1.89) | 3.96 (1.46)
  Postoperative week 12 | 6.69 (2.23) | 4.38 (1.92)
Statistical Analysis 1: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Diqufosol vs Hyaluronate; Linear mixed model was used to compare measurement data between the 2 groups by considering the correlation between both eyes of each patient at postoperative week 4; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Diqufosol vs Hyaluronate; Linear mixed model was used to compare measurement data between the 2 groups by considering the correlation between both eyes of each patient at postoperative week 12; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

5. Primary Outcome: Corneal Fluorescein Staining That is Related to Dry Eye Severity.
Description: Ocular surface damage was assessed by the National Eye Institute (NEI) workshop grading system, and corneal fluorescein staining was evaluated. Instillation of fluorescein in both eyes. After 1 or 2 full blinks, the intensity of staining of both cornea was scored. According to the National Eye Institute (NEI) workshop grading system, the cornea was divided into five sections. The minimum staining score was 0 and the maximum staining score was 15 points (up to 3 points for each section).
  0 : best score (no corneal damage) 15 : worst score (severe corneal damages)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores
Units Other Than Participants: eyes
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 30 | 33
Number analyzed (eyes) | 45 | 49
scores
  Baseline | 1.52 (0.41) | 1.78 (0.28)
  Postoperative week 1 | 2.09 (0.45) | 2.88 (0.31)
  Postoperative week 4 | 1.09 (0.33) | 1.73 (0.23)
  Postoperative week 12 | 0.48 (0.77) | 1.21 (1.45)
Statistical Analysis 1: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis

6. Primary Outcome: Lissamine Green (LG) Conjunctival Staining That is Related to Dry Eye Severity
Description: Ocular surface damage was assessed by the National Eye Institute (NEI) workshop grading system, and conjunctival LG staining were evaluated. Instillation of 1% lissamine green in both eyes. After 1 or 2 full blinks, the intensity of staining of both medial and lateral bulbar conjunctiva was cored. According to the National Eye Institute (NEI) workshop grading system, the conjunctiva was divided into six sections. The minimum staining score was 0 and the maximum staining score was 18 points (up to 3 points for each section).
  0 : best score (no conjunctival damage) 18 : worst score (severe conjunctival damages)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: eyes
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 30 | 33
Number analyzed (eyes) | 45 | 49
Scores on a scale
  Baseline | 1.40 (0.32) | 1.91 (0.22)
  Postoperative week 1 | 2.56 (0.73) | 3.86 (0.50)
  Postoperative week 4 | 0.86 (1.18) | 2.31 (2.12)
  Postoperative week 12 | 0.36 (0.76) | 1.33 (2.04)
Statistical Analysis 1: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis
Statistical Analysis 3: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis

7. Secondary Outcome: Grades of Anterior Chamber Cells.
Description: Anterior chamber inflammation was examined with a slit-lamp clinically, and divided into six grades using the Standardization of Uveitis Nomenclature (SUN) working group grading scheme.
  grade 0 : <1 cell in field, grade 0.5 : 1-5 cells in field, grade 1 : 6-15 cells in field, grade 2 : 16-25 cells in field grade 3 : 26-50 cells in field, grade 4 : >50 cells in field Field size is a 1 mm X 1 mm slit beam
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: grade
Units Other Than Participants: eyes
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 30 | 33
Number analyzed (eyes) | 45 | 49
grade
  Baseline | 0 (0) | 0 (0)
  Postoperative week 1 | 1.54 (0.34) | 1.78 (0.25)
  Postoperative week 4 | 0.16 (0.26) | 0.36 (0.22)
  Postoperative week 12 | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: Diqufosol vs Hyaluronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.151, Mixed Models Analysis

8. Secondary Outcome: Number of Participants Who Stop Using the Eye Drops Due to Drug-related Discomfort
Description: Drug-related discomfort is defined as having started after eye drop instillation and lasting several minutes, occurring every time during instillation at any time up to 12 weeks into the follow-up period. Patients that had any adverse events or wanted to stop using the eye drops were excluded from the study, but these patients were included in the safety evaluation.
Time Frame: 12 weeks
Population: Overall, 1 of 31 patients (3.22%), a 64-year-old man who underwent bilateral sequential same-day cataract surgery, stopped using the study eye drops owing to severe irritation in the D group.
Measure: Number; unit: participants
Arm/Group | Diqufosol | Hyaluronate
Number analyzed (Participants) | 31 | 33
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Patients that had any adverse events or wanted to stop using the eye drops were excluded from the study, but these patients were included in the safety evaluation.
Arm/Group | Diqufosol | Hyaluronate
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 1/31 | 0/33
OTHER ADVERSE EVENTS (reported when occurring in more than 3.23% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diqufosol (N=31) | Hyaluronate (N=33)
Severe irritation (Eye disorders) | 1 (1) | 0 (0) — 64-year-old man who underwent bilateral sequential same-day cataract surgery, stopped using the study eye drops owing to severe irritation in the D group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No